CLINICAL TRIAL: NCT03438448
Title: Perioperative Myocardial Ischemia: Implementation of Troponin Monitoring, Economic Analysis and Further Insights Into Pathophysiology
Brief Title: Perioperative Myocardial Ischemia: Troponin Monitoring,Cost-effectiveness, Insights Into Pathophysiology
Acronym: PMI
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-IMP-2015-95
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Ischemia; Myocardial Injury; Morality
Keywords: Ultrasensitive Troponin T; MINS; Cost-effectiveness; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High sensitive Troponin T monitoring — Three determinations of Roche high-sensitive troponin T (99th percentile (14 ng/L) for each patient: preoperative (during the preoperative visit or just before surgery), 48h, and 72h after surgery. If a rise and/or fall of hs-cTnT with at least one value above the 99th percentile upper reference is detected, a clinical evaluation and a 12-lead ECG will be performed. If no ECG changes, ischemic symptoms, or pulmonary edema to fulfill the diagnostic for PMI the patients will undergo an echocardiographic study.

SUMMARY:
Background: Despite preoperative screening, technical improvements and increased patient monitoring, perioperative myocardial infarction (PMI) remains the first cause of morbidity and mortality within 30 days after surgery. Moreover, the available evidence indicates worrying rise of risk in postoperative patients with only elevated troponins reflecting cardiac injury, but without a conventional clinical diagnosis of myocardial infarction according to current definition. Worldwide, annually approximately 300 million adults undergo major non cardiac surgery and 10 million of them are estimated to suffer a myocardial injury after non-cardiac surgery (MINS), defined as a prognostically relevant increase of a troponin T peak of 0.03 ng/ml or greater. Many of the patients with MINS does not fulfill the universal definition of myocardial infarction, rarely experience ischemic symptoms and their prognosis is very poor (1 out of 10 die at 30 days).Troponin levels needed to be monitored in order to MINS diagnose and high sensitive cardiac troponin T assays are currently the most frequently used.

Methods: Patients with high cardiovascular risk undergoing major non-cardiac surgery will be selected from the daily surgical program during a two years period Three determinations of hs-cTnT for each patient will be obtained. The proportion of patients with MINS and pre- and post-operative thresholds of hs-cTnT that would be prognostically relevant will be determined. The cost-effectiveness analysis of hs-cTnT monitoring compared with usual care will be undertaken. Finally using computed tomography angiography (CTA) and cardiac magnetic resonance imaging (MRI) pathophysiology of MINS will be determined, whether is due to plaque rupture, supply-demand mismatch, non-ischemic cardiac cause or non-cardiac cause.

Discussion: The study will evaluate the feasibility and impact of implementing the hs-cTnT monitoring program in the Hospital de la Santa Creu i Sant Pau of Barcelona, as well as its cost-effectiveness. Moreover, this is the first study which will determine pre and postoperative thresholds of hs-cTnT and with minimally invasive diagnostic tools will evaluate potential mechanisms involved in perioperative ischemic events.

DETAILED DESCRIPTION:
The study consists of four sub studies

* Troponin monitoring implementation - Sub study A
* Preoperative and postoperative hs-cTnT threshold - Sub study B
* Economic analysis - Sub study C
* Advanced cardiac imaging case-control study - Sub study D

Study A:To implement and evaluate a Troponin T monitoring program in patients with high cardiovascular risk undergoing major non-cardiac surgery, the investigators will include prospectively patients with one or more of the following inclusion criteria (intervention cohort). Age, sex, type of surgery, revised cardiac risk index, history of coronary artery disease, history of cardiac arrest, history of congestive heart failure, history of peripheral vascular disease, history of stroke, history of a transient ischemic attack, chronic renal failure, history of deep venous thrombosis or pulmonary embolism, diabetes, hypertension, current atrial fibrillation, chronic obstructive pulmonary disease, type of treatment (statins and antithrombotic treatments) will be collected.

The investigators will obtain three determinations of Roche high-sensitive troponin T (99th percentile (14 ng/L) for each patient: preoperative (during the preoperative visit or just before surgery), 48h, and 72h after surgery. If a rise and/or fall of hs-cTnT with at least one value above the 99th percentile upper reference is detected, a clinical evaluation and a 12-lead ECG will be performed. If no ECG changes, ischemic symptoms, or pulmonary edema to fulfill the diagnostic for PMI the patients will undergo an echocardiographic study.

Study B: All patients included in study A (see above) will included. The investigators will measure high sensitivity cardiac troponin T using a Roche Elecsys 2010 analyzer (limit of detection 5.0 ng/L, 99th percentile 14 ng/L, a 10% coefficient of variation at 13 ng/L) at three predefined time points: preoperatively (during the preoperative visit or just before surgery), at 48h and 72h after surgery. The main outcome will be 30 day and 1 year mortality.

Study C: To analyze the cost-effectiveness of a hs-cTnT screening program for the detection of PMI compared to the current practice (no screening). The investigators will structure a model as a decision tree analysis. Two alternatives will be considered: the application of screening program for detection of PMI versus current practice, based on the application of standard treatments in the presence of ischemic symptoms.

Study D: All the patients from hs-cTnT screening study mentioned above (A) who fulfill MINS criteria will be recruited in this study. After obtaining written informed consent, all variables included risk factors, comorbidities, medical treatment and perioperative data will be recollected by researchers. Within the postoperative hospitalization period, CTA and MRI studies will be performed in all cases.

Two groups of patients will be distinguished :

* MINS/PMI group: composed by patients with hs-cTnT value higher than 50% of preoperative level, without symptoms, without ECG changes related to ischemia, neither new wall abnormalities in the postoperative echocardiogram. Moreover PMI group will be composed by patients with perioperative myocardial infarction according the current definition.
* Control group: composed by patients without PMI or MINS.

After a matching analyses for the principal confounding factors (age, sex, Lee index, type of surgery), one control for each case will be selected to complete CTA and MRI examinations.

In MRIs the investigators will do an analysis of global and segmental contractility baseline perfusion, a pharmacological stress with adenosine, and an assessment of necrosis and myocardial viability by studying late gadolinium enhancement contrast. In CTAs the investigators will evaluate plaque morphology, plaque size and composition, stenosis and remodeling index.

Given these findings, and with the information provided by clinical history and eventual ECG changes, the investigators will classify MINS patients as (1) due to plaque rupture, (2) supply-demand mismatch, (3) non-ischemic cardiac cause, or (4) non-cardiac cause.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 65 years.
* Age < 65 years and documented cardiovascular disease (history of coronary artery disease, history of congestive heart disease, history of stroke, history of peripheral vascular disease).
* Renal insufficiency (GF <60ml/min).

Exclusion criteria:

Patients undergoing non cardiac surgery that do not require an overnight hospital admission or that only receive infiltrative (i.e., local) or topical anesthesia.

Ages: 45 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥ 65 years or < 65 years with documented cardiovascular disease (history of coronary artery disease, history of congestive heart disease, history of stroke, history of peripheral vascular disease) undergoing a major non-cardiac surgery can considered for eligibility. Eligible Patients will be approached for informed consent after surgery and before hospital discharge.
Sampling Method: Probability Sample
Enrollment: 1510 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 month and 1 year after surgery
  Occurence of all cause mortality

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 month and 1 year after surgery
  Occurrence of MACE: myocardial infarction, unstable angina, congestive heart failure, new atrial fibrillation, stroke or pulmonary embolism
Medication modifications | 1 month and 1 year after surgery
  Starting new medication or modifying dose

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Alonso-Coello, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- HospitalSCSP, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alvarez-Garcia J, Popova E, Vives-Borras M, de Nadal M, Ordonez-Llanos J, Rivas-Lasarte M, Moustafa AH, Sole-Gonzalez E, Paniagua-Iglesias P, Garcia-Moll X, Vilades-Medel D, Leta-Petracca R, Oristrell G, Zamora J, Ferreira-Gonzalez I, Alonso-Coello P, Carreras-Costa F. Myocardial injury after major non-cardiac surgery evaluated with advanced cardiac imaging: a pilot study. BMC Cardiovasc Disord. 2023 Feb 10;23(1):78. doi: 10.1186/s12872-023-03065-6. PMID 36765313
- [Derived] Popova E, Alonso-Coello P, Alvarez-Garcia J, Paniagua-Iglesias P, Rue-Monne M, Vives-Borras M, Font-Gual A, Gich-Saladich I, Martinez-Bru C, Ordonez-Llanos J, Carles-Lavila M. Cost-effectiveness of a high-sensitivity cardiac troponin T systematic screening strategy compared with usual care to identify patients with peri-operative myocardial injury after major noncardiac surgery. Eur J Anaesthesiol. 2023 Mar 1;40(3):179-189. doi: 10.1097/EJA.0000000000001793. Epub 2023 Jan 11. PMID 36722187